CLINICAL TRIAL: NCT06200662
Title: Pain Relief in Premature Newborns Through Maternal Intervention During Venipuncture: Effectiveness, Experiences of Parents and Carers
Brief Title: Pain Relief in Premature Newborns Through Maternal Intervention During Venipuncture
Acronym: PREMAMANDOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 8836
Record Dates: First submitted 2023-08-29; First posted 2024-01-11 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2023-08

CONDITIONS: Premature Newborns

STUDY DESIGN:
Intervention Model Description: This is a single-centre crossover study which plans t o include up to 48 newborns (objective: 40 analysable subjects, visit S and visit M carried out) for whom two different analgesic strategies will be applied, each at one of the two time points of the crossover:
  * a control treatment, referred to here as treatment S: standard and recommended non- pharmacological analgesic strategies carried out by the carer alone
  * an experimental treatment, referred to here as treatment M: overall non-pharmacological analgesic strategies carried out by the mother The groups are therefore the "order S then M" group and the "order M then S" group.
  The order of visits was determined randomly (prior randomisation) for each mother-child dyad.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- premature newborns (Other): premature newborns . 2 groups composed of the same children but benefiting from 2 different analgesic strategies, each applied at one of two different times. The groups compared were the "order S then M" group and the "order M then S" group.
  Interventions: Other: Analgesic strategies during the S visit:; Other: Analgesic strategies at visit M
- premature (Other): premature newborns . 2 groups composed of the same children but benefiting from 2 different analgesic strategies, each applied at one of two different times. The groups compared were the "order S then M" group and the "order M then S" group.
  Interventions: Other: Analgesic strategies during the S visit:; Other: Analgesic strategies at visit M

INTERVENTIONS:
Other: Analgesic strategies during the S visit: — Analgesic strategies during the S visit: standard and recommended non-pharmacological analgesic strategies used by the CRI: administration of sugar solution, support for non-nutritive sucking with a dummy and wrapping in a nappy.
Other: Analgesic strategies at visit M — Analgesic strategies at visit M: overall non-pharmacological analgesic strategies carried out by the mother: sucking on a sugar solution, supporting non-nutritive sucking with a dummy, contact, etc.

SUMMARY:
Extremely premature newborn infants (ELNs) admitted to hospital are exposed to stressful and painful stimuli, and often to maternal separation, which can affect their long-term neurological development. Child- and family-centred developmental care (CFDC) in neonatology aims to adapt the hospital environment to the needs of the child, support the continued presence of the family and help to improve their future.

Specific assessment and appropriate analgesic treatment are therefore priorities for preserving the well-being and cerebral development of this population, which is particularly vulnerable to pain. Pain relief for certain procedures necessary for the care of newborn babies, such as venipuncture (PV), remains inadequate. Venipuncture is a common procedure in the first few weeks of life for very premature newborns. Its analgesic treatment is based on non-medicinal strategies largely carried out in the nurse's own role: non-nutritive suctioning combined with the administration of a sugar solution and wrapping. In line with the SDCEF philosophy, and reinforced by the "zero separation" concept, parental involvement in the treatment of their newborn's pain becomes natural and fundamental. A number of studies have shown the benefits of parents' presence and participation through specific isolated analgesic actions. Skin- to-skin contact (PAP) is one of these and has multiple benefits for the newborn. However, in practice, when a PV is necessary for a very premature baby, its use as a pain-relieving strategy is hampered by a number of obstacles. As NN are naturally oriented towards the maternal voice, using it is a new approach to analgesia. In an innovative study carried out in a single centre, direct maternal voice contact, in addition to the usual non- pharmacological analgesic strategies, reduced the NN's pain, without completely eliminating it during heel sampling (a skin incision known to be more painful than a PV). This analgesic strategy should therefore be combined with other non-pharmacological strategies, taking advantage of all maternal skills.

DETAILED DESCRIPTION:
* Information visit (V0 - 1 day): parents are informed by the clinical research nurse (CRN);
* Inclusion visit (V0): inclusion, collection of consent from the 2 holders of parental authority, collection of anamnestic data by the CRI;
* Visit S and visit M (V0 to ≤ 7 d): random order, installation of the NN in a room dedicated to recordings, analgesic strategies (see below), performance at each visit of a PV (necessary for care) by the IRC, collection of behavioural data by video sequences centred on the NN's face.

Analgesic strategies during the S visit: standard and recommended non-pharmacological analgesic strategies used by the CRI: administration of sugar solution, support for non-nutritive sucking with a dummy and wrapping in a nappy.

Analgesic strategies at visit M: overall non-pharmacological analgesic strategies carried out by the mother: sucking on a sugar solution, supporting non-nutritive sucking with a dummy, contact, etc.

direct voice (from 5 minutes before to 5 min after PV), wrap in a nappy and manual, and offer to grasp the finger.

Analysis of behavioural data: NFCS scores obtained from analysis of video sequences by 10 s periods (basal, per and post stimulation) by 2 blind assessors on the type of analgesia used (carer or mother).

ELIGIBILITY:
Inclusion Criteria:

* Very premature babies born before the gestational age (GA) of 32 weeks of amenorrhoea (SA) whose corrected age (CA) does not exceed 34 SA at the time of their participation.
* NN requiring close biological monitoring by a PV.
* Hospitalised in the NN medicine and intensive care unit at Strasbourg hospital.
* Consent obtained from both holders of parental authority.
* Person covered by a social health insurance scheme.

Exclusion Criteria:

* Any known malformation affecting one or more organs.
* Cerebral lesions discovered o n cerebral ultrasound (intraventricular haemorrhage grade > 2, periventricular leukomalacia).
* Unstable clinical state as judged by the investigator and the medical team.
* Transfer to another hospital centre expected before the end of the study period.

  * Mother: Minor. Deprived of liberty by judicial or administrative decision. Under legal protection. Severe psychological pathology. Drug addiction. Difficulty understanding and/or reading the language.

French.

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
NFCS (Neonatal Facial Coding System) | 7 days
  the NFCS pain score assessed during a PV in two conditions:
  * maternal absence: "carer" analgesia (visit S) ;
  * maternal involvement: "mum" pain (M visit). This is a validated 4-item scale describing facial mimics in NN. The analysis was based on video sequences and blinded to the type of analgesia used. The possible score is from 0 to 4 and will be binarised to a value of "1"; the primary endpoint (PEC) is therefore the proportion of neonates with a score of "1". greater than or equal to 1.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie RABATEL, Principal Investigator — Médecine et Réanimation du Nouveau-né Hôpital de Hautepierre CHU de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, Bas-Rhin, France